CLINICAL TRIAL: NCT06244381
Title: NUTRITIONAL OPTIMIZATION IN THE DIFFERENT PHASES OF CRITICAL ILLNESS. Comparison of the Urea/Creatinine Ratio With Indirect Calorimetry.
Brief Title: Indirect Calorimetry Versus Urea-creatinine Ratio to Evaluate Catabolism in Critically Ill Patients
Status: Completed | Type: Observational
Sponsor: Hospital Sao Domingos (Other)
Responsible Party: Principal Investigator, José Raimundo Araujo de Azevedo, Clinical Researcher, Hospital Sao Domingos
Other Study IDs: hsd0124
Record Dates: First submitted 2024-01-29; First posted 2024-02-06 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Critically Ill
Keywords: Catabolism; Indirect calorimetry; Urea/creatinine ratio; Critically ill; COVID-19
MeSH Terms: conditions — Critical Illness; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to evaluate the efficiency of the urea/creatinine ratio as a catabolism marker compared to indirect calorimetry to optimize nutritional support in critically ill patients.

DETAILED DESCRIPTION:
The most recent ESPEN guideline on nutritional support in critically ill patients identifies 3 phases in the evolution of critically ill patients: the early acute phase (formerly EBB Phase), characterized by endogenous energy production and activation of autophagy that limits full caloric-protein intake; the late period of the acute phase, when endogenous energy production has reduced to a basal level and autophagy is no longer manifested, and the late or rehabilitation phase. The identification of each of these moments is not based on precise elements. Despite this division into phases, there is no clear evidence of metabolic behavior, especially in the second and third phases, when the catabolic state gives way to anabolism.

Currently, monitoring catabolism is complicated since there is no available biomarker with acceptable sensitivity and specificity. 3-methyl histidine and nitrogen balance are not available in everyday life. As catabolism is not measured, its presence and severity only become apparent when muscle loss and weakness set in.

Recently, Haines et al., analyzing a population of patients with persistent severe disease, who are patients with prolonged hospitalization and with no resolution in the ICU, showed that continued catabolism is their metabolic hallmark and was measured by the urea/creatinine ratio persistently high.

The phases of severe illness could then be defined based on the UCR relationship. The ratio must be high in the early acute and late acute phases and may be a marker of the beginning of the late phase of recovery and anabolism.

Indirect calorimetry, the gold standard for determining energy expenditure energy, has revealed in studies that it can be the marker of the beginning of the anabolic when energy expenditure increases rapidly. This behavior of indirect calorimetry was observed in COVID-19 but has also been demonstrated in other patient populations.

Although indirect calorimetry can represent a reliable measure for determining the beginning of the anabolic phase, it is not a widely available measurement in ICUs, unlike urea and creatinine measurements that are part of routine daily exams in ICUs.

The urea/creatinine ratio may be an efficient catabolism marker to guide nutritional therapy in critically ill patients. Evidence to confirm this hypothesis can be obtained by comparing the urea/creatinine ratio with indirect calorimetry, which is the gold standard for evaluating energy expenditure and catabolism in these patients.

The primary objective will be to correlate the behavior of the urea/creatinine ratio with the energetic expenditure measured by indirect calorimetry in patients with severe forms of COVID-19 to identify the beginning of the anabolic phase that would be translated by a reduction in UCR and an increase in energy expenditure in IC. Secondarily, correlate other catabolism markers with calorimetry results. They are serum albumin, hemoglobin, and C-reactive protein.

ELIGIBILITY:
Inclusion Criteria: Adult patients with severe COVID-19 submitted to determination of energetic expenditure between the first and twentieth day of ICU stay -

Exclusion Criteria: patients who, upon arrival at the hospital, had a serum creatinine level above 4.0 mg°/dL, chronic kidney disease patients undergoing dialysis, and patients undergoing dialysis treatment during their stay in the ICU.

-

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Twenty critically ill COVID-19 patients admitted to a 35-bed ICU intended for patients with COVID-19 from April to August 2021 and who underwent determination of energy expenditure with indirect calorimetry on days 1, 4, 7, 9, 14, 17, and 20 days after admission, and who did not have serum creatinine > 4.0 mg/dL upon admission, were not chronic dialysis patients and did not undergo dialysis treatment during the study period. The urea, creatinine, C-reactive protein, hemoglobin, and albumin results will be obtained from the hospital's electronic medical record during the study period.
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
Urea/creatinine ratio | 30 days
  Compare urea/creatinine ratio with indirect calorimetry to determine catabolism and optimize nutritional support in critically ill COVID-19 patients.

SECONDARY OUTCOMES:
Serum albumin | 30 days
  Compare albumin with indirect calorimetry to determine catabolism and optimize nutritional support in critically ill COVID-19 patients.
Hemoglobin concentration | 30 days
  Compare hemoglobin concentration with indirect calorimetry to determine catabolism and optimize nutritional support in critically ill COVID-19 patients.
C-reactive protein | 30 days
  Compare C-reactive protein with indirect calorimetry to determine catabolism and optimize nutritional support in critically ill COVID-19 patients.

CONTACTS AND LOCATIONS:
Overall Officials: JOSE AZEVEDO, MD, PhD, Study Director — Hospital São Domingos
Locations (1):
- Hospital Sao Domingos, São Luiz, Maranhão, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Singer P, Blaser AR, Berger MM, Calder PC, Casaer M, Hiesmayr M, Mayer K, Montejo-Gonzalez JC, Pichard C, Preiser JC, Szczeklik W, van Zanten ARH, Bischoff SC. ESPEN practical and partially revised guideline: Clinical nutrition in the intensive care unit. Clin Nutr. 2023 Sep;42(9):1671-1689. doi: 10.1016/j.clnu.2023.07.011. Epub 2023 Jul 15. PMID 37517372
- [Result] Long CL, Dillard DR, Bodzin JH, Geiger JW, Blakemore WS. Validity of 3-methylhistidine excretion as an indicator of skeletal muscle protein breakdown in humans. Metabolism. 1988 Sep;37(9):844-9. doi: 10.1016/0026-0495(88)90118-7. PMID 3138511
- [Result] Haines RW, Zolfaghari P, Wan Y, Pearse RM, Puthucheary Z, Prowle JR. Elevated urea-to-creatinine ratio provides a biochemical signature of muscle catabolism and persistent critical illness after major trauma. Intensive Care Med. 2019 Dec;45(12):1718-1731. doi: 10.1007/s00134-019-05760-5. Epub 2019 Sep 17. PMID 31531715
- [Result] Niederer LE, Miller H, Haines KL, Molinger J, Whittle J, MacLeod DB, McClave SA, Wischmeyer PE. Prolonged progressive hypermetabolism during COVID-19 hospitalization undetected by common predictive energy equations. Clin Nutr ESPEN. 2021 Oct;45:341-350. doi: 10.1016/j.clnesp.2021.07.021. Epub 2021 Aug 3. PMID 34620338
- [Result] Long CL, Schaffel N, Geiger JW, Schiller WR, Blakemore WS. Metabolic response to injury and illness: estimation of energy and protein needs from indirect calorimetry and nitrogen balance. JPEN J Parenter Enteral Nutr. 1979 Nov-Dec;3(6):452-6. doi: 10.1177/014860717900300609. PMID 575168
- [Result] Monk DN, Plank LD, Franch-Arcas G, Finn PJ, Streat SJ, Hill GL. Sequential changes in the metabolic response in critically injured patients during the first 25 days after blunt trauma. Ann Surg. 1996 Apr;223(4):395-405. doi: 10.1097/00000658-199604000-00008. PMID 8633918